CLINICAL TRIAL: NCT03437629
Title: Influences of Different Temporary Cement on Retention Rate and Dental Sensitivity of Temporary Crown on Vital Teeth - Randomized Clinical Trial
Brief Title: Influences of Different Temporary Cement on Retention Rate of Temporary Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.294.913
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: MTA; Calcium Hydroxide; Dental Crown

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide temporary cement (Active Comparator): Cementation of a temporary crown with cement based on calcium hydroxide.
  Interventions: Procedure: Temporary cement based on Calcium Hydroxide
- MTA temporary cement (Active Comparator): Cementation of a temporary crown with cement based on Mineral trioxide aggregate .
  Interventions: Procedure: MTA temporary cement

INTERVENTIONS:
Procedure: Temporary cement based on Calcium Hydroxide — Confection of a temporary crown with acrylic resin; Finishing and polishing; relative isolation with cotton and gauze; Manipulation of the temporary cement based on Calcium Hydroxide; Cement insertion on the internal surface of the temporary crown; Excess cement removal; Occlusal Adjustment.
  Arms: Calcium Hydroxide temporary cement
Procedure: MTA temporary cement — Confection of a temporary crown with acrylic resin; Finishing and polishing; relative isolation with cotton and gauze; Manipulation of the temporary cement based on Mineral trioxide aggregate; Cement insertion on the internal surface of the temporary crown; Excess cement removal; Occlusal Adjustment.
  Arms: MTA temporary cement

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, split-mouth, evaluate the success rate (retention rate and dental sensibility) of temporary dental crown cemented on vital teeth. The composition of the cement (Based on calcium hydroxide; and based on mineral trioxide aggregate) will be evaluated. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
The confecction of temporary prosthesis is a fundamental step in the prosthetic process of definitive total crowns. The temporary cementation should provide sufficient retention between the intervals of the consultations, be biocompatible and not present high solubility. The aim of this study is through a randomized clinical trial, double blind, splithmouth, evaluate the success rate (retention rate and dental sensibility) of temporary dental crown cemented on vital teeth. The composition of the cement (Based on calcium hydroxide; and based on mineral trioxide aggregate) will be evaluated. Twenty participants with at least two vital teeth with the need to confection of definitive total crowns (each participant) will be selected who present. The teeth will be randomly divided into 2 different groups according to the temporary cement composition (Based on calcium hydroxide; and based on mineral trioxide aggregate). Data will be collected, tabulated and submitted to statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers; both genres; presence of at least two teeth with indication of total crowns; good oral hygiene.

Exclusion Criteria:

* Dentures or orthodontics; presence of periodontal disease and,or parafunctional habits; systemic disease and, or severe psychological; constant use of analgesic and, or anti-inflammatory or allergic response to dental products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate (retention rate and absence of sensibility) of temporary dental crown cemented with different temporary cement with a 6 months follow up | 6 mounths

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Jabbari YS, Al-Rasheed A, Smith JW, Iacopino AM. An indirect technique for assuring simplicity and marginal integrity of provisional restorations during full mouth rehabilitation. Saudi Dent J. 2013 Jan;25(1):39-42. doi: 10.1016/j.sdentj.2012.10.003. Epub 2012 Nov 10. PMID 23960554
- [Background] Arora SJ, Arora A, Upadhyaya V, Jain S. Comparative evaluation of marginal leakage of provisional crowns cemented with different temporary luting cements: In vitro study. J Indian Prosthodont Soc. 2016 Jan-Mar;16(1):42-8. doi: 10.4103/0972-4052.164911. PMID 27134427
- [Background] da Rosa WLO, Cocco AR, Silva TMD, Mesquita LC, Galarca AD, Silva AFD, Piva E. Current trends and future perspectives of dental pulp capping materials: A systematic review. J Biomed Mater Res B Appl Biomater. 2018 Apr;106(3):1358-1368. doi: 10.1002/jbm.b.33934. Epub 2017 May 31. PMID 28561919
- [Background] Hill EE, Lott J. A clinically focused discussion of luting materials. Aust Dent J. 2011 Jun;56 Suppl 1:67-76. doi: 10.1111/j.1834-7819.2010.01297.x. PMID 21564117
- [Background] Malkoc MA, DemIr N, Sengun A, Bozkurt SB, Hakki SS. Cytotoxicity of temporary cements on bovine dental pulp-derived cells (bDPCs) using realtime cell analysis. J Adv Prosthodont. 2015 Feb;7(1):21-6. doi: 10.4047/jap.2015.7.1.21. Epub 2015 Feb 17. PMID 25722833
- [Background] von Arx T. [Mineral trioxide aggregate (MTA) a success story in apical surgery]. Swiss Dent J. 2016;126(6):573-95. doi: 10.61872/sdj-2016-06-02. French, German. PMID 27377433